CLINICAL TRIAL: NCT00119587
Title: A Double-Blind, Randomized, Comparative Study of Darbepoetin Alfa Given Once Weekly or Once Every Other Week for Treatment of Anemia in Hemodialysis Subjects
Brief Title: Darbepoetin Alfa Treatment of Anemia in Hemodialysis Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Global Development Leader, Amgen Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20010219
Record Dates: First submitted 2005-06-30; First posted 2005-07-14 (Estimated); Last update posted 2007-12-28 (Estimated); Status verified 2007-12

CONDITIONS: Anemia
Keywords: Hemodialysis; darbepoetin alfa; Clinical Trial; Amgen
MeSH Terms: conditions — Anemia | interventions — Darbepoetin alfa

INTERVENTIONS:
Drug: darbepoetin alfa

SUMMARY:
The purpose of this study is to compare once a week and once every other week darbepoetin alfa on the change in hemoglobin levels between the screening/baseline period and the evaluation period (weeks 25-30). This study will also assess the change in mean hemoglobin over 4 week intervals, instability of hemoglobin concentrations, darbepoetin alfa dosing requirements and red blood cell transfusions.

ELIGIBILITY:
Inclusion Criteria: - -Receiving hemodialysis for at least 6 months before screening - -Clinically stable as judged by the investigator - Stable IV rHuEPO therapy administered 1, 2 or 3 times per week for at least 8 weeks before screening (stable is defined as less than or equal to 25% change [up or down] in weekly dose and no change in frequency over 8 weeks) - Adequate iron stores (serum ferritin greater than or equal to 100μg/L) during the screening period - Available for follow up assessments - Before any study specific procedure is carried out, the subject, or his/her legally acceptable representative must give informed consent for participation in the study Exclusion Criteria: - -Treatment for grand mal epilepsy in the last 6 months - Congestive heart failure (New York Heart Association [NYHA] class III or IV)- - Uncontrolled hypertension, defined as a predialysis diastolic blood pressure measurement greater than or equal to 110mmHg during the screening period - Clinical evidence of current uncontrolled hyperparathyroidism (e.g., serum parathyroid hormone greater than 1500pg/mL) within the past 12 months - Major surgery within 3 months before screening (excludes vascular access surgery) - Previously diagnosed HIV or chronic hepatitis B infection - Clinical evidence of current malignancy excluding basal cell or squamous cell carcinoma of the skin - Systemic hematological disease (e.g., sickle cell anemia, myelodysplastic syndromes, hematological malignancy); myeloma; hemolytic anemia - Alanine transaminase (ALT) and aspartate transaminase (AST) greater than 2 times the upper limit of the normal range - RBC transfusion(s) within 12 weeks before screening or during the screening/baseline period, or active bleeding - Clinical evidence of current systemic infections - Androgen therapy within 12 weeks before screening - No prior treatment with darbepoetin alfa - Currently enrolled in, or has not yet completed a period of at least 30 days since ending, other investigational device or drug trial(s). Subjects receiving other investigational agent(s) may only enter the study after discussion and agreement with Amgen - Pregnancy (women of child-bearing potential must be using adequate contraception) - Breast feeding - Psychiatric, addictive, or other disorder that compromises ability to give truly informed consent or is likely to alter compliance - Anticipating or scheduled for a living-related kidney transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-08; Study Completion 2003-09

PRIMARY OUTCOMES:
Comparison between once a week and once every other week darbepoetin alfa on the change in Hb level between the screening/baseline period and the evaluation period (weeks 25-30)

SECONDARY OUTCOMES:
Instability of Hb concentration during the evaluation period
Weekly dose and frequency of darbepoetin alfa during the evaluation period
RBC transfusions during the evaluation period.

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com